CLINICAL TRIAL: NCT00825682
Title: The Effect of Reflexology on Radiation-related Fatigue and QOL in Breast Cancer Patients: a Pilot Study.
Brief Title: The Effect of Reflexology on Radiation-related Fatigue in Breast Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Dorit Gamus, Director, Complementary Medicine Service, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-07-4923-DG-CTIL
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-10

CONDITIONS: Fatigue
Keywords: Breast cancer; Radiation therapy; Reflexology; Fatigue; Quality of life; Sleep disturbance
MeSH Terms: conditions — Fatigue; Breast Neoplasms; Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 20 breast cancer patients scheduled for adjunctive radiation treatment will be recruited for this study to receive reflexology treatment initiated at the beginning of radiation therapy, once a week, for 10 weeks.
  Interventions: Other: Reflexology treatment.
- 2 (No Intervention): 20 breast cancer patients, scheduled for adjunctive radiation treatment, matched by age to the intervention group will receive treatment as usual, and will be evaluated by the same measures as the intervention group.

INTERVENTIONS:
Other: Reflexology treatment. — Reflexology treatments (45 min. each) will be initiated at the beginning of radiation therapy, once a week, for 10 weeks.The treatment includes manual pressure on specific points of foot soles and massage of the calf area, adapted individually to each patient.
  Other Names: Foot massage
  Arms: 1

SUMMARY:
Oncologic patients often report increased fatigue during and after radiation therapy. Reflexology treatment has been demonstrated to alleviate symptoms of fatigue, nausea, and anxiety in oncologic patients treated with chemotherapy. The aim of the study is to evaluate the effect of reflexology on fatigue, quality of life, and quality of sleep of breast cancer patients during and after radiation therapy.

DETAILED DESCRIPTION:
Reflexology (foot massage) is a complementary medicine technique which is performed by manual pressure on specific areas of the feet. Reflexology is based on a system of zones and reflex areas that are believed to reflect an image of the body on the feet with a premise that such work effects a physical change to the body.

The effect of reflexology on fatigue, quality of life, and quality of sleep of 20 breast cancer patients during and after radiation therapy will be compared to age-matched control group of 20 breast cancer patients treated by radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer adult patients scheduled to receive adjuvant radiation therapy

Exclusion Criteria:

* Open wounds or evidence of metastases on the lower limbs
* Touch therapy or other complementary therapy other than intervention procedure

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-05; Primary Completion 2009-02 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorit D Gamus, MD, PhD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Hospital,, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deng G, Cassileth BR, Yeung KS. Complementary therapies for cancer-related symptoms. J Support Oncol. 2004 Sep-Oct;2(5):419-26; discussion 427-9. PMID 15524070
- [Background] Kohara H, Miyauchi T, Suehiro Y, Ueoka H, Takeyama H, Morita T. Combined modality treatment of aromatherapy, footsoak, and reflexology relieves fatigue in patients with cancer. J Palliat Med. 2004 Dec;7(6):791-6. doi: 10.1089/jpm.2004.7.791. PMID 15684846
- [Background] Yang JH. [The effects of foot reflexology on nausea, vomiting and fatigue of breast cancer patients undergoing chemotherapy]. Taehan Kanho Hakhoe Chi. 2005 Feb;35(1):177-85. doi: 10.4040/jkan.2005.35.1.177. Korean. PMID 15778569
- [Background] Cassileth BR, Vickers AJ. Massage therapy for symptom control: outcome study at a major cancer center. J Pain Symptom Manage. 2004 Sep;28(3):244-9. doi: 10.1016/j.jpainsymman.2003.12.016. PMID 15336336
- [Background] Quattrin R, Zanini A, Buchini S, Turello D, Annunziata MA, Vidotti C, Colombatti A, Brusaferro S. Use of reflexology foot massage to reduce anxiety in hospitalized cancer patients in chemotherapy treatment: methodology and outcomes. J Nurs Manag. 2006 Mar;14(2):96-105. doi: 10.1111/j.1365-2934.2006.00557.x. PMID 16487421

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included 72 breast cancer patients, scheduled for complementary radiation therapy at the Cancer Center at Tel Hashomer Hospital during the years 2008-2011. Participants were recruited to the experimental and control groups, on a voluntary basis.
Pre-assignment Details: Exclusion criteria: breast cancer patients with metastatic lesions on lower limbs, coagulation disorders and patients receiving other contact treatments.
Groups:
- Reflexology Group: The experimental group included 47 women with breast cancer scheduled for adjunctive radiation treatment. The women received reflexology treatment initiated at the beginning of radiation therapy, once a week (45 min each), for 10 weeks.
- Control Group: The control group (no intervention,treatment as usual)included 25 breast cancer patients, scheduled for adjunctive radiation treatment, who completed the same questionnaires at the same time points as the as the intervention group.
Period: Overall Study
Arm/Group | Reflexology Group | Control Group
Started | 47 | 25
Completed | 34 | 20
Not Completed | 13 | 5
Not completed — personal reasons/ inconvenience | 13 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reflexology Group | Control Group | Total
Number analyzed (Participants) | 47 | 25 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 22 | 61
  >=65 years | 8 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (9.47) | 52.3 (11.78) | 54.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 25 | 72
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Israel | 47 | 25 | 72

OUTCOME MEASURES:

1. Primary Outcome: The Lee Fatigue Scale
Description: The Lee Fatigue Scale consists of 18 items related to fatigue and energy: 13 items in the fatigue subscale and 5 items in the energy subscale. The mean of the 13 items in the fatigue subscale (range from 0-10) and the mean of the 5 items in the energy subscale (range from 0-10) are calculated. Higher scores indicate higher levels of perceived fatigue and energy . Items in the energy subscale were recoded, and a Lee fatigue total score was calculated as the average of all 18 items (ranging between 0 and 10), higher scores indicating higher levels of fatigue.
  The Cronbach's Alpha reliability coefficient of the English version of the questionnaire is 0.77 . The questionnaire's validity and reliability have been established in cancer patients.
Time Frame: Beginning of study (initiation of radiation therapy and reflexology), 5 weeks after start (end of radiation therapy), 10 weeks after start
Population: The final analysis included 33 women in the experimental group and 20 in the control group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Reflexology Group | Control Group
Number analyzed (Participants) | 33 | 20
units on a scale
  begining of the study | 3.71 (1.76) | 3.68 (1.56)
  5 weeks | 3.9 (1.57) | 5.32 (1.61)
  10 weeks | 3.6 (1.45) | 4.52 (2.05)

2. Secondary Outcome: The Multidimensional Quality of Life Scale Cancer MQOLS-CA Was Written by Padilla (1992) and Translated Into Hebrew by Dorit Pud (2007).
Description: The questionnaire includes 33 items describing different forms in which the disease may affect patient's quality of life. For each item, subjects are asked to mark the number that best describes their feelings right now, in a Likert scale ranging between 0 and 10. Items include happiness feelings, anxiety levels, how affected are the social ties because of the disease, etc.
  A total quality of life score was calculated as the average of all 33 items (ranging between 0 and 10), higher scores indicating a better quality of life.
Time Frame: as for outcome 1
Population: The final ananlysis included 34 women in the experimental group, and 20 women in the control group.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Reflexology Group: The experimental group included 47 women with breast cancer scheduled for adjunctive radiation treatment. The women received reflexology treatment initiated at the beginning of radiation therapy, once a week (45 min each), for 10 weeks. Five women did not begin the study and 8 women did not complete reflexology treatments due to personal reasons / inconvenience
Arm/Group | Reflexology Group | Control Group
Number analyzed (Participants) | 34 | 20
Scores on a scale
  beginning of study | 4.23 (1.36) | 4.09 (1.13)
  5 weeks | 4.17 (1.25) | 4.58 (1.09)
  10 weeks | 4.04 (1.25) | 4.49 (1.02)

3. Secondary Outcome: The General Sleep Disturbance Scale (GSDS), Compiled by Lee (1992) and Translated Into Hebrew by Dr. Dorit Pud (2007)
Description: examines several aspects of sleep disorders and includes 21 items that describe feelings and behaviors associated with sleep during the last week. It uses a 0 (never) to 7 (every day) Likert scale on questions like feeling nervous during the day; falling asleep while unplanned and using sleeping pills.
  A total sleep disturbance score was calculated as the average of all 21 items (ranging between 0 and 7), higher scores indicating a worse outcome.
Time Frame: as for outcome 1
Population: The final analysis included 34 women in the experimental group and 20 in the control group.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Reflexology Group | Control Group
Number analyzed (Participants) | 34 | 20
Scores on a scale
  beginning of study | 2.51 (1.02) | 2.35 (0.84)
  5 weeks | 2.27 (0.67) | 2.67 (0.86)
  10 weeks | 2.19 (0.73) | 2.49 (0.87)

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: no adverse effects were reported during the study
Arm/Group | Reflexology Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/25
Other Adverse Events (participants affected / at risk) | 0/47 | 0/25

LIMITATIONS AND CAVEATS:
This was a pilot non-randomized controlled study, with a relatively small sample and a single therapist.The control group received no additional intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No